CLINICAL TRIAL: NCT04469660
Title: Impact of COVID-19 Pandemic on the Psychological Wellbeing of Healthcare
Brief Title: Impact of COVID-19 Pandemic on the Psychological Wellbeing of Healthcare Professionals in India
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Max Healthcare Insititute Limited (Other)
Responsible Party: Sponsor
Other Study IDs: Onco Survey_COVID-19
Record Dates: First submitted 2020-07-13; First posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Psychological Stress
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To Study the epidemiology of psychological distress among healthcare professionals of Max Super Speciality Hospital,Saket ,New Delhi in India during the COVID-19 Pandemic and assess the implications for providing psychological interventions(or therapeutic services)

DETAILED DESCRIPTION:
To Study the epidemiology of psychological distress among healthcare professionals of Max Super Speciality Hospital,Saket ,New Delhi in India during the COVID-19 Pandemic and assess the implications for providing psychological interventions(or therapeutic services).

Hypothesis: There is likelihood of psychological distress impacting healthcare professionals' mental well-being as a result of their role in the healthcare setup during the COVID-19 pandemic. Study design-The questionnaire assessing the psychological wellbeing shall be administered via digital means of communication to healthcare professionals and support staff (doctors, nurses, paramedics, front office and support staff) across Max Super Speciality Hospital, Saket, New Delhi that currently employs 1295 individuals in the current category.

Participation in the study will be voluntary and informed consent will be sought prior to the survey administration. Participants' responses will remain anonymous, with an assurance of confidentiality.

ELIGIBILITY:
Inclusion Criteria Healthcare professionals working in Max Super Speciality Hospital Saket New Delhi Healthcare professionals inclusive of doctors, nurses paramedics front office employee and support staff Healthcare professionals above 18 years of age Healthcare professionals residing in India

Exclusion Criteria Non-employees of Max Super Speciality Hospital Saket New Delh Healthcare professionals residing outside India

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthcare Professionals of Max Super Speciality Hospital,Saket,New Delhi
Sampling Method: Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2020-05-18 (Actual); Primary Completion 2020-08-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Therapeutic Sessions emphasizing on Stress | 3 Months
  The therapeutic sessions will emphasize on aspects of anxiety, depression, grief, post traumatic impact, loss, fear and so on, using standardized therapeutic techniques of psychotherapy. If the individual is in need of further management or somatic symptom related treatment, they will be guided for pharmacotherapy.

SECONDARY OUTCOMES:
Resilience building and planning | 3 Months
  Resilience building and planning will be implemented via individual, group and/or online based training portals to the cohort falling in the range of mild-moderate levels of psychological distress.

CONTACTS AND LOCATIONS:
Overall Officials: Hiba Siddiqui, Principal Investigator — Max Super Speciality Hospital,Saket,New Delhi
Locations (1):
- Max Super Speciality Hospital Saket, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided
Yet not decided